CLINICAL TRIAL: NCT01169376
Title: Therapeutically Applicable Research to Generate Effective Treatments (TARGET) for Neuroblastoma
Brief Title: Biomarkers in Young Patients With Neuroblastoma
Status: Completed | Type: Observational
Sponsor: Children's Oncology Group (Network)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Other Study IDs: ANBL10B1; COG-ANBL10B1 (Other: Children's Oncology Group); CDR0000681912 (Other: Clinical Trials.gov); NCI-2011-02246 (Registry Identifier: CTRP (Clinical Trial Reporting Program))
Record Dates: First submitted 2010-07-23; First posted 2010-07-26 (Estimated); Last update posted 2016-05-18 (Estimated); Status verified 2016-05

CONDITIONS: Neuroblastoma
Keywords: disseminated neuroblastoma; localized resectable neuroblastoma; localized unresectable neuroblastoma; regional neuroblastoma; stage 4S neuroblastoma
MeSH Terms: conditions — Neuroblastoma | interventions — DNA Methylation; Comparative Genomic Hybridization; Amplified Fragment Length Polymorphism Analysis

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No

INTERVENTIONS:
Genetic: DNA analysis
Genetic: DNA methylation analysis
Genetic: RNA analysis
Genetic: comparative genomic hybridization
Genetic: mutation analysis
Genetic: polymorphism analysis

SUMMARY:
RATIONALE: Studying samples of tumor tissue from patients with cancer in the laboratory may help doctors identify and learn more about biomarkers related to cancer.

PURPOSE: This research study is studying biomarkers in young patients with neuroblastoma.

DETAILED DESCRIPTION:
OBJECTIVES:

Primary

* To discover the therapeutically relevant driver mutations in high-risk pediatric neuroblastoma.

Secondary

* To identify a set of highly annotated neuroblastoma specimens (primary tumors and cell lines) for comprehensive genomic analyses, validation studies, resequencing efforts, and future functional assays.
* To define genome-wide DNA copy number and allelic status in at least 300 high-risk and 50 low-risk neuroblastoma primary untreated tumors, and 30 human neuroblastoma-derived cell lines.
* To define the genome-wide methylation profile of neuroblastoma in a minimum of 200 high-risk cases.
* To define the genome-wide microRNA expression profile of neuroblastoma in a minimum of 200 high-risk cases.
* To define genome-wide RNA expression signatures, including splice variations, in the same tumors and cell lines studied above.
* To identify mutations in candidate therapeutic targets using a staged resequencing strategy with ultimate genome-scale next generation resequencing of 3 genomes for 200 high-risk cases: the neuroblastoma genome and transcriptome as well as the paired constitutional genome.
* To characterize the relapsed high-risk neuroblastoma genome and epigenome.

OUTLINE: This is a multicenter study.

Previously collected samples are analyzed to define the genome-wide DNA copy number and allelic status; to define the genome-wide methylation profile of high-risk neuroblastoma cases; to define the genome-wide microRNA expression profile of high-risk neuroblastoma cases; to define the genome-wide RNA expression and relating gene expression to DNA copy number and gene polymorphisms, DNA methylation, and microRNA expression; to resequence three genomes: the neuroblastoma genome, the transcriptome, and the paired constitutional genome; and to characterize the relapsed high-risk neuroblastoma genome and epigenome.

PROJECTED ACCRUAL: A total of 300 tumor samples from patients with high-risk disease, 50 tumor samples from patients with low-risk primary neuroblastoma, and 30 human neuroblastoma-derived cell lines will be accrued for this study.

ELIGIBILITY:
DISEASE CHARACTERISTICS:

* Registered on the COG-ANBL00B1 Neuroblastoma Biology Study or its CCG or POG precursor
* Sufficient high-quality tumor material available for the proposed studies meeting the following criteria:

  * Tissue histopathologic review with > 70% tumor cells in sections adjacent to areas used for nucleic acid preparation
  * Matched normal cells (blood or uninvolved bone marrow) available
  * ≥ 5 μg DNA available
  * ≥ 5 μg RNA available
  * ≥ 200 mg tissue available
* Tumor samples must meet 1 of the following criteria:

  * High-risk tumor

    * With or without MYCN amplification
    * With or without tumor progression or relapse (during ≥ 2.5 years of follow up)
    * Patients aged 18 months to 5 years
  * Low-risk tumor

    * Primary neuroblastoma
    * Stage I disease (completely resected)
    * No event in ≥ 3 years of follow up
  * Cell lines representing diverse high-risk genetics including with or without MYCN amplification and clinical course (at diagnosis or after relapse)

PATIENT CHARACTERISTICS:

* Not specified

PRIOR CONCURRENT THERAPY:

* Not specified

Max Age: 30 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Study Population: Patients registered on the COG-ANBL00B1 Neuroblastoma Biology Study
Sampling Method: Non-Probability Sample
Enrollment: 380 (Estimated)
Dates: Start 2010-07; Primary Completion 2016-05 (Actual); Study Completion 2016-05 (Actual)

PRIMARY OUTCOMES:
Discovery of therapeutically relevant driver mutations

SECONDARY OUTCOMES:
Identification of a set of neuroblastoma specimens for analyses
Genome-wide DNA copy number and allelic status
Genome-wide methylation profile
Genome-wide microRNA expression profile
Genome-wide RNA expression signatures
Identification of mutations in candidate therapeutic targets
Characterization of the relapsed high-risk neuroblastoma genome and epigenome

CONTACTS AND LOCATIONS:
Overall Officials: John M. Maris, MD, Principal Investigator — Children's Hospital of Philadelphia